CLINICAL TRIAL: NCT00190996
Title: The Safety and Effectiveness of Duloxetine Compared With Placebo and Its Long-Term Safety and Efficacy in the Treatment of Predominant Stress Urinary Incontinence
Brief Title: Evaluate Safety and Efficacy of Duloxetine in Predominant Stress Urinary Incontinence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8049; F1J-EW-SBCC
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-01-26 (Estimated); Status verified 2007-01

CONDITIONS: Urinary Incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Duloxetine Hydrochloride
Drug: placebo

SUMMARY:
The purposes of this study are to determine whether duloxetine can help subjects with stress urinary incontinence and to see whether the effects of duloxetine can be maintained.

ELIGIBILITY:
Inclusion Criteria:

* Female diagnosed with stress urinary incontinence

Exclusion Criteria:

* Currently taking a monoamine oxidase inhibitor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2765
Dates: Start 2003-01; Study Completion 2006-06

PRIMARY OUTCOMES:
Assess the efficacy of Duloxetine compared with placebo in women with predominant stress urinary incontinence as measured by a reduction in incontinent episode frequency.

SECONDARY OUTCOMES:
Evaluate the maintenance of effect on IEF in long-term use
Kings Health Questionnaire
Patient Global Impression of Improvement Questionnaire
Safety effects

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey, United Kingdom

REFERENCES:
- [Derived] Cardozo L, Lange R, Voss S, Beardsworth A, Manning M, Viktrup L, Zhao YD. Short- and long-term efficacy and safety of duloxetine in women with predominant stress urinary incontinence. Curr Med Res Opin. 2010 Feb;26(2):253-61. doi: 10.1185/03007990903438295. PMID 19929591